CLINICAL TRIAL: NCT02062918
Title: Effectiveness of Abdominal Belt for the Chronic Low Back Pain Treatment
Brief Title: Abdominal Belt Use to Treat Low Back Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Jamil Natour, Head of Rheumatology Division, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CEP?UNIFESP-1726/10
Record Dates: First submitted 2014-02-12; First posted 2014-02-14 (Estimated); Last update posted 2014-02-14 (Estimated); Status verified 2014-02

CONDITIONS: Chronic Low Back Pain
Keywords: Abdominal belt; Chronic low back pain; Pain; Functional capacity
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control group (No Intervention): Patients in the control group did not use an abdominal belt.
- Experimental group (Experimental): Patients were instructed in how to use the abdominal belt for activities of physical effort that exacerbated lumbar pain as well as during moments of pain, and not to use it during rest. They should record the number of hours of belt use per day on spreadsheets distributed for this purpose.
  Interventions: Device: Abdominal belt

INTERVENTIONS:
Device: Abdominal belt
  Arms: Experimental group

SUMMARY:
Objectives: To assess the effectiveness of an abdominal belt in the treatment of chronic mechanical-postural low back pain.

Methods: A randomized controlled trial was carried out, involving 60 consecutively selected patients with chronic low back pain randomly allocated to an intervention group (use of abdominal belt) and control group (non-use of abdominal belt). Patients were evaluated at the baseline of the study (T0) as well as 1 (T1), 3 (T3) and 6 months (T6) after the inclusion. The patients were assessed for: pain (VAS); functional capacity (Roland Morris), patient satisfaction (Likert scale); and number of anti-inflammatory pills ingested. Intention-to-treat analysis was also used.

Hypothesis - abdominal belt will improve pain in chronic low back pain patients

ELIGIBILITY:
Inclusion Criteria:

* patients from both genders,
* between 18 and 65 years of age,
* who sought medical care for a complaint of lumbar pain,
* diagnosed with Chronic low back pain, with VAS for pain between 4 and 8 cm (0-10),
* who agreed to participate in the study and signed terms of informed consent.

Exclusion Criteria:

* diagnosis or under diagnostic investigation of low back pain from secondary causes (spondyloarthopathy, infection, neoplasm, complete sciatica),
* fibromyalgia,
* previous spinal surgery,
* litigation (patients on leave from work or in work leave processes due to low back pain);
* having changed physical activity in previous three months;
* body mass index (BMI) higher than 30;
* acupuncture treatment or physiotherapy in the previous three months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2010-01; Primary Completion 2010-03 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Change in pain using VAS | Baseline, after 1,3, and 6 months

SECONDARY OUTCOMES:
Change in functional capacity (Roland-Morris questionnaire) | Baseline, after 1,3 and 6 months
Change in hours of abdominal belt use | Baseline, after 1,3 and 6 months
Change in patient satisfaction with treatment using VAS | Baseline, after 1,3 and 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Universidade Federal de Sao Paulo, São Paulo, São Paulo, Brazil